CLINICAL TRIAL: NCT05154487
Title: Phase 2 Study of Alpelisib and Fulvestrant for PIK3CA-mutated Estrogen Receptor (ER)-positive Endometrioid Endometrial Cancers
Brief Title: A Study of Alpelisib and Fulvestrant to Treat Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-3069
Record Dates: First submitted 2021-11-23; First posted 2021-12-13 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Endometroid Endometrial Cancer
Keywords: advanced; persistent; recurrent; PIK3CA-mutated; ER-postive
MeSH Terms: conditions — Recurrence | interventions — Alpelisib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apelisib and Fulvestrant (Experimental): alpelisib 300mg orally daily of each 28-day cycle fulvestrant 500mg IM on Day 1 and Day 15 of Cycle 1, then 500mg IM on Day 1 of each 28-day cycle.
  Interventions: Drug: Alpelisib Pill; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: Alpelisib Pill — Kinase inhibitor
  Other Names: Piqray
Drug: Fulvestrant injection — estrogen receptor agonist
  Other Names: Faslodex

SUMMARY:
This is a 2 stage multi-center study designed to evaluate the efficacy of the combination of alpelisib and fulvestrant in patients with PIK3CA-mutated ER-positive endometrioid endometrial cancers by estimating the objective response rate (ORR). Treatment will continue until either unacceptable toxicity, progression of disease, or investigator/patient request for withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have advanced (FIGO 2014 Stage III or IV), persistent, or recurrent endometrial carcinoma, which is not likely to be curable by surgery or radiotherapy. Histologic confirmation of recurrent disease is required. For cases of persistent disease, histologic confirmation of the primary disease with radiologic evidence of progression is required.
2. Patients must have endometrioid histology (all grades allowed) based on hysterectomy or biopsy specimen and have positive expression of ER and oncogenic PIK3CA mutation per criteria below.

   a. PIK3CA mutations considered oncogenic or likely oncogenic. i. Oncogenic/likely oncogenic PIK3CA mutations identified on tests performed by the labs listed on https://ecog-acrin.org/nci-match-eay131-designated-labs will be considered confirmed for the purposes of this study.

   ii. Oncogenic/likely oncogenic PIK3CA mutations identified by other tests will need to be confirmed by the study prior to enrollment.

   b. Estrogen receptor (ER) status will be considered positive if ≥1% of tumor cells demonstrate positive nuclear staining by immunohistochemistry. Pathology report documenting ER status must be provided at enrollment.

   Sites are required to report results of previous MMR and/or MSI status testing in the EDC if available.
3. All patients must have measurable disease. Measurable disease is defined by RECIST version 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be greater than or equal to 10mm when measured by CT, MRI or caliper measurement by clinical exam; or greater than or equal to 20mm when measured by chest x-ray. Lymph nodes must be greater than or equal to 15mm in short axis when measured by CT or MRI.

   Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
4. Prior chemotherapy in the adjuvant setting for Stage I, II, or III or metastatic/recurrent/Stage IV is permitted. Prior chemoradiotherapy for a pelvic recurrence is permitted.

   Prior immunotherapy and/or targeted therapy is allowed in addition to, in combination with, in lieu of, or subsequent to prior chemotherapy.

   Prior hormone therapy (progesterone, tamoxifen, aromatase inhibitor) is allowed and not considered a prior line of therapy. Prior treatment with fulvestrant not allowed.

   There are no limits on the number of prior lines of chemotherapy. Patients who received prior chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade less than or equal to 1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to enrollment. A washout period of at least 21 days is required between last chemotherapy dose and initiation of therapy.

   Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and initiation of therapy.
5. Patient must be able to swallow oral medications.
6. Patient must have an ECOG performance status of 0 to 2.
7. Patients must have adequate glucose control as defined by the following (both criteria must be met):

   * Fasting blood glucose (FBG) ≤140/dL (7.7mmol/L) AND
   * Hemoglobin A1c (HbA1c) ≤6.4%
8. Patients must have adequate organ and marrow function as defined below NOTE: Institutional/laboratory upper limit of normal = ULN Institutional/laboratory lower limit of normal = LLN

   Bone marrow function:
   * Absolute neutrophil count (ANC) greater than or equal to 1000/mcl
   * Platelets greater than or equal to 100,000 cells/mcl
   * Hemoglobin greater than or equal to 8 g/dL (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after erythrocyte transfusion).

   Renal function:

   • Creatinine Clearance ≥ 35 mL/min using Cockcroft-Gault formula

   Pancreatic function:
   * Fasting Serum amylase ≤ 2 × ULN
   * Fasting Serum lipase ≤ ULN

   Hepatic function:
   * Bilirubin less than or equal to 1.5 x ULN (Patients with Gilbert's syndrome with a total bilirubin ≤2 times ULN and direct bilirubin within normal limits are permitted).
   * ALT (alanine aminotransferase) and AST (aspartate aminotransferase) less than or equal to 3 x ULN
   * Albumin greater than or equal to 2.8 g/dL
9. Patients must have signed an approved informed consent and authorization permitting release of personal health information.
10. Patients must be at least 18 years of age.
11. Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing a highly effective form of contraception during the study treatment and for 8 weeks after stopping the treatment.

Highly effective contraception methods include combination of any of the following (NOTE: Estrogen containing contraceptives are prohibited):

* Use of oral, injected, or implanted hormonal contraceptives or;
* Placement of an intrauterine device (IUD) or intrauterine system (IUS);
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository;
* Total abstinence or;
* Male/female sterilization. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to registration. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.

Exclusion Criteria:

1. Patients who have previously received fulvestrant or any PIK3CA, PI3K, mTOR, or AKT inhibitor.
2. Patients with clear cell, serous, carcinosarcoma, mixed histology endometrial cancers, or uterine sarcomas.
3. Patients with known intolerance or hypersensitivity to alpelisib or fulvestrant, or any of their excipients.
4. Patient has had major surgery within 14 days prior to study treatment start and/or has not recovered from major side effects.
5. Patients with an established diagnosis of diabetes mellitus type I or uncontrolled type II (based on fasting blood glucose [FBG] and HemoglobinA1c [HbA1c], see inclusion criterion 67).
6. Patients with history of osteonecrosis of the jaw.
7. Patients with concomitant invasive malignancy or a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the past five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol.
8. Patients with active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment, fungal infection, or detectable viral infection (such as known human immunodeficiency virus (HIV) positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]). Screening is not required for enrollment.
9. Patients with a serious pre-existing medical condition(s) that would preclude participation in this study (for example: interstitial lung disease or pneumonitis, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment (i.e. estimated creatinine clearance <30ml/min), history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or pre-existing chronic condition resulting in baseline grade 2 or higher diarrhea).
10. Patients with a known history of cardiac disease. This includes:

    * Uncontrolled hypertension, defined as systolic greater than 150mm Hg or diastolic greater than 90mm Hg despite antihypertensive medications
    * Myocardial infarction, unstable angina, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to registration.
    * New York Heart Association (NYHA) Class II or greater congestive heart failure.
    * History of clinically significant cardiac arrhythmias (i.e. ventricular tachycardia or ventricular fibrillation, complete left bundle branch block, high grade AV block (e.g. bifascicular block, Mobitz type II and third degree AV block without pacemaker in place) or serious cardiac arrhythmia requiring medication. This does not include asymptomatic atrial fibrillation with controlled ventricular rate.
    * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or Fridericia QT correction formula (QTcF) > 470 msec at screening.
    * Cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) within 6 months prior to the first date of study therapy.
    * Syncope of cardiovascular etiology,
    * Sudden cardiac arrest.
11. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to the start of the treatment:

    * Strong CYP3A4 inducers
    * Inhibitors of BCRP.
12. Patients who are pregnant or breast-feeding.
13. Patients with known central nervous system metastases which was not previously treated and not fulfilling the following 3 criteria to be eligible for the study:

    * Completed prior therapy (including radiation and/or surgery) for CNS metastases ≥ 28 days prior to the start of study entry and
    * CNS tumor is clinically stable at the time of screening and
    * Participant is not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases.
14. Patients with an impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study drugs (i.e. ulcerative disease; uncontrolled nausea, vomiting and/or diarrhea; malabsorption syndrome; clinical signs and symptoms of gastrointestinal obstruction; and/or patients who require parenteral hydration and/or nutrition).
15. Patients who plan to receive live attenuated vaccines within 1 week of start of alpelisib and during the study. Patients should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG< yellow fever, varicella, and TY21a typhoid vaccines.
16. Patients with active bleeding or pathologic conditions that carry high risk of bleeding such as known bleeding disorder or coagulopathy.
17. Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 30 days prior to dosing, or within 5 half-lives of the investigational product, whichever is longer.
18. Patient is not able to understand and to comply with study instructions and requirements, including oral administration of study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | Response to treatment is assessed by RECIST Version 1.1 criteria every 8 weeks with CT scan or MRI through completion of treatment (complete or partial response). Patients receive treatment until disease progression and are followed for 5 years.
  To determine the objective response rate of the combination of alpelisib and fulvestrant in patients with advanced, persistent or recurrent PIK3CA-mutated ER-positive endometrioid endometrial cancer. Respnse criteria based on RECIST Version 1.1 (complete or partial response).

SECONDARY OUTCOMES:
Drug Toxicity (Side Effects) | Side effects are monitor from the start of treatment to discontinuation of treatment assessed every 4 weeks. Patients are treated until disease progression and are followed for 5 years.
  Drug toxicity will be assessed by collecting adverse event data every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gaillard, MD, Study Chair — GOG Foundation
Locations (11):
- United States (11):
  - City of Hope, Duarte, California
  - AdventHealth Gynecologic Oncology, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Ascension St. Vincent, Indianapolis, Indiana
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Kettering Health Cancer Center, Kettering, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Legacy Good Samaritan Medical Center, Portland, Oregon
  - Legacy Meridian Park Medical Center, Tualatin, Oregon
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided